CLINICAL TRIAL: NCT02751073
Title: Evaluation of Vaginal and Urinary Microbiome Markers as Predictors of Post-Surgical Urinary Tract Infection
Brief Title: Evaluation of the Relationship Between Vaginal and Lower Urinary Tract Microbiomes and Infection After Hysterectomy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John A. Occhino, Assistant Professor of Obstetrics-Gynecology, Mayo Clinic
Other Study IDs: 15-006300
Record Dates: First submitted 2016-02-22; First posted 2016-04-26 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Pelvic Organ Prolapse; Hysterectomy; Urinary Tract Infection
Keywords: Microbiota; Proteome
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal swabs and urine samples (catheterized and clean-catch) collected longitudinally throughout the perioperative period.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn more about the microbes (bacteria) that live in the vagina and the bladder. The investigators are doing this research study to understand the relationship between microbes (the microbiome) and the occurrence of urinary tract infection following surgical removal of the uterus and pelvic organ prolapse repair. The investigators expect Lactobacillus and Gardnerella will be the dominant organisms for most women. Non-Lactobacillus dominant microbiome communities will be more common in women who ultimately develop postoperative urinary tract infection.

DETAILED DESCRIPTION:
The goal of this pilot study is to characterize the presence and stability of the microbial community in the vagina and lower urinary tract in a cohort of 20 postmenopausal women undergoing transvaginal hysterectomy with pelvic reconstruction for pelvic organ prolapse. The investigators intend to collect longitudinal samples in the preoperative, intraoperative, and postoperative time period in order to understand the pervasiveness of the microbes in the vagina and lower urinary tract, and to identify, in a very preliminary way, particular microbes that may be associated with postoperative urinary tract infection.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females (defined by cessation of menses for one full year)
* Planned surgical correction of pelvic organ prolapse with transvaginal hysterectomy and concomitant pelvic reconstruction for uterovaginal prolapse
* Scheduled surgery date within 4 weeks of study consent
* Physically able to self-collect vaginal swabs and clean-catch urine samples

Exclusion Criteria:

* Women who are premenopausal, pregnant or nursing
* Currently taking or have taken antibiotics in the past 2 weeks
* History of recurrent urinary tract infections
* History of mesh complications, including erosion/extrusion
* Non-vaginal approach to hysterectomy or prolapse repair

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women undergoing pelvic reconstructive surgery for pelvic organ prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05-31 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Identification of baseline vaginal microbiome through DNA extraction and 16S rRNA gene sequencing | 1 day (Pre-operative Urogynecology surgical consultation visit)
  Vaginal swabs will be collected from participants at the surgical consultation visit. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the vagina.
Identification of baseline urinary tract microbiome through DNA extraction and 16S rRNA gene sequencing | 1 day (Pre-operative Urogynecology surgical consultation visit)
  Urine sample will be collected from participants at the surgical consultation visit. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the urinary tract.
Identification of pre-operative vaginal microbiome through DNA extraction and 16S rRNA gene sequencing | Within 4 weeks of baseline sample collected at Urogynecology surgical consultation visit)
  Vaginal swabs will be collected from participants on the day of surgery, prior to entering the surgical suite. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the vagina.
Identification of pre-operative urinary tract microbiome through DNA extraction and 16S rRNA gene sequencing | Within 4 weeks of baseline sample collected at Urogynecology surgical consultation visit)
  Urine sample will be collected from participants on the day of surgery, prior to entering the surgical suite. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the urinary tract.
Identification of the immediate postoperative vaginal microbiome through DNA extraction and 16S rRNA gene sequencing | Within 6 hours of collecting the pre-operative sample
  Vaginal swabs will be collected from participants at the end of the surgical procedure. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the vagina.
Identification of the immediate postoperative urinary tract microbiome through DNA extraction and 16S rRNA gene sequencing | Within 6 hours of collecting the pre-operative sample
  Urine sample will be collected from participants at the end of the surgical procedure. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the urinary tract.
Identification of the postoperative vaginal microbiome through DNA extraction and 16S rRNA gene sequencing | 12-18 hours after surgery
  Vaginal swabs will be collected from participants the morning following surgery, after removal of the vaginal packing. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the vagina.
Identification of the postoperative urinary tract microbiome through DNA extraction and 16S rRNA gene sequencing | 12-18 hours after surgery
  Urine sample will be collected from participants the morning following surgery, after removal of the vaginal packing. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the urinary tract.
Identification of vaginal microbiome in the setting of postoperative urinary tract infection through DNA extraction and 16S rRNA gene sequencing | Within the first 6 weeks after surgery
  Vaginal swabs will be collected at the onset of symptomatic urinary tract infection during the time period between hospital dismissal and 6-week postoperative surgical visit. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition in the vagina in the setting of urinary tract infection and compare to microbiome of vagina during the perioperative period.
Identification of urinary tract microbiome in the setting of postoperative urinary tract infection through DNA extraction and 16S rRNA gene sequencing | Within the first 6 weeks after surgery
  Urine sample will be collected at the onset of symptomatic urinary tract infection during the time period between hospital dismissal and 6-week postoperative surgical visit. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the urinary tract in the setting of urinary tract infection and compare to microbiome of the urinary tract during the perioperative period.
Identification of key biomarkers associated with risk of postoperative urinary tract infection through proteomic mass spectrometry analysis of vaginal swab collected in the setting of postoperative urinary tract infection | Within the first 6 weeks after surgery
  Vaginal swab collected at onset of symptomatic urinary tract infection during the time period between hospital dismissal and 6-week postoperative surgical visit. Proteomic mass spectrometry analysis of vaginal swab will be conducted. The investigators will use this proteomic information together with the microbial community identified with 16S rRNA to identify a transition point or key biomarkers associated with risk of postoperative urinary tract infection.
Identification of the vaginal microbiome at least 6 weeks following surgery through DNA extraction and 16S rRNA gene sequencing | 6 weeks (up to 8 weeks)
  Vaginal swabs will be collected from participants at the Urogynecology post-surgical consultation. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the vagina.
Identification of the postoperative urinary tract microbiome at least 6 weeks following surgery through DNA extraction and 16S rRNA gene sequencing | 6 weeks (up to 8 weeks)
  Urine sample will be collected from participants at the Urogynecology post-surgical consultation. DNA extraction and 16S rRNA gene sequencing undertaken to analyze the microbial community composition of the urinary tract.

CONTACTS AND LOCATIONS:
Overall Officials: John A Occhino, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Occhino JA, Byrnes JN, Wu PY, Chen J, Walther-Antonio MR. Preoperative vaginal microbiome as a predictor of postoperative urinary tract infection. Sci Rep. 2024 Nov 22;14(1):28990. doi: 10.1038/s41598-024-78809-1. PMID 39578602